CLINICAL TRIAL: NCT03199378
Title: Neuropsychological Norms for Ethnically Diverse Florida Elders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: Mayo Clinic (Other); Mt. Sinai Medical Center, Miami (Other); Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: FloridaElderNorms
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Caucasian: English speaking Caucasian individuals
  Interventions: Other: Neuropsychological Testing
- African American: English speaking African American individuals
  Interventions: Other: Neuropsychological Testing
- Hispanic: Spanish speaking Hispanic individuals
  Interventions: Other: Neuropsychological Testing

INTERVENTIONS:
Other: Neuropsychological Testing — Each group will be administered a battery of neuropsychological tests

SUMMARY:
The goal of this proposal is to collect normative data from a sample of ethnically diverse Florida elders on a brief, standardized neuropsychological test battery . The norms collected in this multi-cultural dataset will provide appropriate corrections for demographic and sociocultural variables that contribute to performance variance on neuropsychological tests. By accounting for these variables, the normative corrections will improve specificity and eliminate disparities in diagnostic validity and clinical utility of neuropsychological tests when administered to Florida's ethnic minority elders.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or above.
* Any gender.
* Primary language of English or Spanish.
* Self-identifies as Hispanic, non-Hispanic Black/African American, or non-Hispanic Caucasian.
* Global Clinical Dementia Rating (CDR) score = 0.

Exclusion Criteria:

* Memory decline reported by participant, informant (if available), or study clinician.
* Currently uncontrolled health condition that could affect cognition.
* Abnormal findings on current neurologic examination.
* History of chronic neurological diseases (stroke, active seizure disorder, parkisonism, TBI with subsequent cognitive change.
* Current substance abuse or history of substance dependence.
* History of chronic psychiatric disease (Bipolar disorder, schizophrenia).
* Currently active mood disorder. History of depression or anxiety is acceptable if symptoms are controlled (Score <6 on the Geriatric Depression Scale). If taking psychoactive mood medication dosage must be stable for at least one month prior to testing.
* Use of cognitive enhancing medications (i.e. cholinesterase inhibitors, memantine).
* Need for assistance in activities of daily living due to cognitive reasons.
* Sensorimotor deficits that would interfere with ability to perform neuropsychological tests.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals in the state of Florida who are over the age of 60 and self-identify as Hispanic, non-Hispanic Black/African American, or non-Hispanic Caucasian.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological norms | 1 year
  Norm referenced scores from the sample population

CONTACTS AND LOCATIONS:
Overall Officials: John Lucas, Ph.D, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mt. Sinai Medical Center, Miami, Florida
  - University of South Florida, Tampa, Florida